CLINICAL TRIAL: NCT02682745
Title: Single Dosing Clinical Trial to Assess the Pharmacokinetic Characteristics and Safety/Tolerability of HL151 Formulation in Healthy Male Subjects
Brief Title: Single Dosing Clinical Trial of HL151
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HL-BPSR-101
Record Dates: First submitted 2016-02-03; First posted 2016-02-15 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Rhinitis, Allergic, Perennial
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- R-T1-T2 (Experimental): First period: administration of reference drug, Second period: administration of test drug l, Third period : administration of test drug ll
  Interventions: Drug: HL151; Drug: TALION tab.
- R-T2-T1 (Experimental): First period : administration of reference drug, Second period : administration of test drug ll, Third period : administration of test drug l
  Interventions: Drug: HL151; Drug: TALION tab.
- T1-T2-R (Experimental): First period : administration of test drug l, Second period : administration of test drug ll, Third period : administration of reference drug
  Interventions: Drug: HL151; Drug: TALION tab.
- T1-R-T2 (Experimental): First period : administration of test drug l, Second period : administration of reference drug, Third period : administration of test drug ll
  Interventions: Drug: HL151; Drug: TALION tab.
- T2-R-T1 (Experimental): First period : administration of test drug ll, Second period : administration of reference drug, Third period : administration of test drug l
  Interventions: Drug: HL151; Drug: TALION tab.
- T2-T1-R (Experimental): First period : administration of test drug ll, Second period : administration of test drug l, Third period : administration of reference drug
  Interventions: Drug: HL151; Drug: TALION tab.

INTERVENTIONS:
Drug: HL151 — Test drug l : HL151, 1T, single oral administration on an empty stomach, Test drug ll : HL151, 1T, single oral administration after meal
Drug: TALION tab. — Reference drug: TALION tab, 1T, every 12 hours, oral administration

SUMMARY:
The purpose of this study is to assess the pharmacokinetic characteristics of bepotastine after single oral administration of TALION tab, a IR formulation of bepotastine as reference drug and HL151, a SR formulation of bepotastine as test drug in healthy male adults. Additionally the safety and tolerability of two drugs will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteer in the age of 19-45
2. Body weight≥50kg and BMI 18~29 kg/m2
3. Subject who sign on an informed consent form willingly

Exclusion Criteria:

1. Subject with serious active cardiovascular, respiratory, hepatologic, renal, hematologic, gastrointestinal, immunologic, dermal, neurologic, or psychological disease or history of such disease
2. Subject with acute disease within 28 days prior to study medication dosing
3. Subject with known for history of disease which affect on the absorption, distribution, metabolism, excretion of drug
4. Subject with clinically significant chronic disease
5. Positive on the test of HBs Ag, anti-HCV Ab, anti-HIV Ab, VDRL
6. Use of any prescription medication within 14 days prior to study medication dosing
7. Use of any medication such as over-the-counter medication including oriental medication within 7 days prior to study medication dosing
8. Subject with clinically significant allergic disease
9. Subject with known for hypersensitivity reaction to bepotastine
10. Subject with any of the following conditions in laboratory test

    * AST/ALT > UNL (upper normal limit) x 2
    * Total bilirubin > UNL x 2
    * Renal failure with CLcr < 50mL/min calculated on Cockcroft-Gault [Cockcroft-Gault GFR = (140-age) * (Wt in kg) / (72 *Cr)]
    * SBP<100mmHg or ≥160mmHg, DBP<60mmHg or ≥100mmHg
    * QTc>440msec on ECG
    * Serum potassium < 3.5 mEq/L or > 5.5 mEq/L
11. Immunological incompetence, immune deficiency or taking immunosuppressants
12. Subject who cannot take standard meal
13. Subject with whole blood donation within 60days, component blood donation within 20days prior to study medication dosing
14. Subject with blood transfusion within 30days prior to study medication dosing
15. Participation in any clinical investigation within 90days prior to study medication dosing
16. Continued excessive use of caffeine (caffeine >five cups/day), alcohol(alcohol>30g/day) and severe heavy smoker(cigarette >10 cigarettes per day)
17. Subject with decision of nonparticipation through investigator's review due to laboratory test results or other excuse such as non-responding to request or instruction by investigator
18. Subject taking inducer or inhibitor of drug metabolism enzyme such as barbital within 30days prior to study medication dosing
19. Subject who are not using adequate means of contraception
20. Subject with genetic problems such as galactose intolerance, Lapp Lactase Deficiency or glucose-galactose malabsorption
21. Subject with history of drug abuse or drug addiction

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2016-02-12 (Actual); Study Completion 2016-02-12 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 24 hours after single administration
Peak Plasma Concentration (Cmax) | 24 hours after single administration

SECONDARY OUTCOMES:
Number of participants with adverse events | Participants will be followed for the duration of study medication dosing days and hospital stay, and follow-up period for maximum 5 days from the discharge

CONTACTS AND LOCATIONS:
Locations (1):
- The Korea Univertisy Anam Hospital, Seoul, South Korea